CLINICAL TRIAL: NCT04426448
Title: The Efficacy, Feasibility, and Acceptability of a Culturally Adapted Brief Intervention for Post-Traumatic Stress Disorder in Severe Mental Illness
Brief Title: Assessment of a Brief Post Traumatic Stress Disorder Intervention for Use in Botswana
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Botswana (Other)
Collaborators: University of KwaZulu (Other)
Responsible Party: Principal Investigator, Keneilwe Molebatsi, Principal Investigator, University of Botswana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBR/RES/IRB/BIO/179
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two equal groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive the BREATHE intervention for three weeks
  Interventions: Behavioral: Brief Relaxation, Education And Trauma HEaling
- Control group (No Intervention): The participants will receive treatment as usual

INTERVENTIONS:
Behavioral: Brief Relaxation, Education And Trauma HEaling — A three-week psychological intervention for PTSD which comprise psychoeducation and breathing retraining to manage anxiety symptoms
  Arms: Intervention group

SUMMARY:
The purpose of this study is to culturally adapt a brief psychological intervention for Post-Traumatic Stress Disorder (PTSD) and assess its efficacy, feasibility, and acceptability in a pilot trial. The intervention has been shown to be efficacious among individuals with comorbid severe mental illness (SMI) and PTSD.

The study will be conducted in three phases. The first phase will determine a description of trauma and responses to traumatic experiences among patients with severe mental illness. The first phase of the study will also determine participants' and mental health care providers' perceptions of suitable PTSD interventions in this middle-income context. The findings will then be used to culturally adapt the brief intervention in the second phase. A pilot trial will be conducted in the third phase of the study.

Participants with comorbid SMI and PTSD will be randomized into two groups (n= 20 intervention group, n= 20 control group). Outcomes of the intervention such as the severity of PTSD symptoms, knowledge about PTSD will be assessed at baseline and at different timelines during the study.

This study will fill the knowledge gap on trauma and its consequences among individuals with severe mental illness in Botswana, it will also contribute to the improvement of clinical practice in the management of PTSD and SMI.

DETAILED DESCRIPTION:
Study participants will be recruited from Sbrana Psychiatric Hospital, the only referral psychiatric hospital in Botswana. The hospital population is representative of the culturally diverse Botswana nation because patients with severe mental illness from the entire country are admitted to the hospital. Forty participants (40) will be recruited and randomized to receive the Brief Relaxation, Education, And Trauma HEaling (BREATHE) intervention or treatment as usual.

The intervention will be delivered by the Principal Investigator who has received training from the intervention developer. Supervision will be provided telephonically.

The BREATHE intervention will be delivered weekly for each participant for a total of three weeks and 4 participants will be enrolled per group resulting in a total of 5 groups. The estimated period of intervention delivery and data collection is therefore expected to last for a period of ~15 weeks.

Outcomes such as anxiety, depressive and PTSD Symptoms, and knowledge about PTSD will be assessed before participants receive the intervention, weekly (following each treatment session), month one and month three after treatment completion. Assessment of feasibility and acceptability will be done at treatment completion with the intervention group. Participants on the control arm will receive outcome measures at the same time points as those receiving the intervention. The investigators will utilize an objective assessment of skin conductance which has been shown to be greater in individuals with PTSD than in individuals without PTSD and similarly increased during a trauma interview in individuals with PTSD compared to individuals who do not have PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand Setswana or English
* The patient must meet the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria for any SMI as categorized for this study (schizophrenia, schizophreniform disorder, schizoaffective disorder, bipolar mood disorder, and severe depressive disorder)
* The patient should meet the criteria for Post-Traumatic Stress Disorder as assessed with the Post Traumatic Checklist-5 (PCL-5)

Exclusion Criteria:

* Currently engaged in psychotherapy for PTSD
* On pharmacotherapy management of PTSD (to control for medication effects on PTSD symptoms)
* Inability to understand informed consent
* Inability to respond to interview questions
* Patients who have suicidal ideation and history of a suicide attempt within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Post Traumatic Checklist-5 | baseline, week 1, 2 ,3,
  Mean Change from Baseline in the severity of PTSD symptoms as assessed with the PCL-5. Total scores for the Post Traumatic Checklist-5 range between 0 and 80 with a cut off score of 33 or higher suggesting the patient may benefit from PTSD treatment. Patients with scores lower than 33 may indicate the patient has sub-threshold symptoms of PTSD
eSense EDA skin conductance device | baseline, week 1, 2 ,3,
  Change in physiological arousal as measured with sensors to assess skin conductance
Mini International Neuropsychiatric Interview (MINI) Plus | baseline, week 3, one month and three months post intervention
  Assessment of symptoms meeting the criteria for PTSD
Consent rates | week 3
  to assess the acceptability of the intervention by dividing the number of participants who meet the criteria for PTSD and meet the inclusion criteria for the pilot trial by the number of those who consent to participate in the trial
Adherence rates | week 3
  to assess acceptability; measured by the total number of sessions attended by the participants and the reasons for non-adherence.
knowledge of PTSD scale (KPTSD) | baseline, week 1, 2 ,3, one month and three months post intervention
  mean difference in the scores obtained in the knowledge of PTSD scale. Higher scores indicate more knowledge of PTSD.
Acceptability of Intervention measure (AIM) | week 3
  Calculation of scores in the Acceptability of Intervention measure. Higher scores indicate greater acceptability
Feasibility of Intervention Measure (FIM) | week 3
  calculation of scores in the Feasibility of Intervention Measure. Higher scores indicate greater feasibility
Patient satisfaction scale | week 3
  calculation of scores in the satisfaction scale. Higher satisfaction with the intervention will be indicated by high scores on the patient satisfaction scale

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | baseline, week 1, 2 ,3, one month and three months post intervention
  Mean Change from Baseline in the severity of depressive symptoms as assessed with the PHQ-9
Clinical Outcomes in Routine Evaluation-Outcome Measure | baseline, week 3, one month and three months post intervention
  Mean difference from Baseline in the severity of psychological distress
Zung self-rating anxiety scale | baseline, week 1, 2 ,3, one month and three months post intervention
  Mean Change from Baseline in the severity of anxiety symptoms as assessed with the Zung anxiety rating scale. Total scores in the Zung self rating scale range from 20 to 80, with scores above 26 indicating severe and extremely severe anxiety.
Post Traumatic Checklist-5 | one month and three months post intervention
  Mean Change from Baseline in the severity of PTSD symptoms as assessed with the Post Traumatic Checklist-5. A five points difference in the total score is an indication that a patient has responded to treatment and 10 points has been determined as a minimum threshold for determining whether the improvement has clinical utility

CONTACTS AND LOCATIONS:
Overall Officials: Keneilwe Molebatsi, MMED (Psych), Principal Investigator — University of Botswana
Locations (1):
- Sbrana Psychiatric Hospital, Lobatse, Botswana

IPD SHARING:
Plan to Share IPD: Yes
The study will be conducted in fulfillment of a Doctor of Philosophy in Psychiatry degree. De-identified data will be shared with the supervisors
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Throughout the study period and one year after completion of write-up
Access Criteria: de-identified coded data will be stored and shared as a statistical package for the social sciences (SPSS) file.

REFERENCES:
- [Derived] Molebatsi K, Ng LC, Chiliza B. A culturally adapted brief intervention for post-traumatic stress disorder in people with severe mental illness in Botswana: protocol for a randomised feasibility trial. Pilot Feasibility Stud. 2021 Sep 3;7(1):170. doi: 10.1186/s40814-021-00904-1. PMID 34479640